CLINICAL TRIAL: NCT04639596
Title: A Randomized Controlled Trial of Mindfulness-based Therapeutic Sailing for Veterans With Psychiatric and/or Substance Use Disorders
Brief Title: Mindfulness-based Therapeutic Sailing (MBTS) Versus Standard Recreation Therapy Activity (SRT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 we never started the study and didn't enroll anyone.
Sponsor: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00122169
Record Dates: First submitted 2020-10-26; First posted 2020-11-20 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Psychiatric Disorder; Substance Use Disorders
Keywords: Psychiatric Disorder; Substance Use Disorders; Sailing; Bowling
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBTS (Experimental): It will consist of four hours of sailing and mindfulness training at the Jordanelle Reservoir. Boats and skippers will be provided by Park City Sailing Association, a non-profit community organization.
  Interventions: Behavioral: Mindfulness-based Therapeutic Sailing (MBTS) versus a standard recreation therapy activity, bowling, (SRT).
- SRT (Experimental): SRT will occur on four separate occasions during the summer of 2019. SRT will consist of 4 hours of bowling at a community bowling alley.
  Interventions: Behavioral: Mindfulness-based Therapeutic Sailing (MBTS) versus a standard recreation therapy activity, bowling, (SRT).

INTERVENTIONS:
Behavioral: Mindfulness-based Therapeutic Sailing (MBTS) versus a standard recreation therapy activity, bowling, (SRT). — This study will be a prospective randomized controlled trial (RCT) of Mindfulness-based Therapeutic Sailing (MBTS) versus a standard recreation therapy activity (bowling) among Veterans with psychiatric and/or substance use disorders.

SUMMARY:
This study will be a prospective randomized controlled trial (RCT) of Mindfulness-based Therapeutic Sailing (MBTS) versus a standard recreation therapy activity (bowling) among Veterans with psychiatric and/or substance use disorders.

The specific aims of this investigation are to determine whether:

1. MBTS will result in greater pre- to post-intervention increases in psychological flexibility and state mindfulness than a standard recreation therapy activity (SRT).
2. MBTS participants will experience greater enjoyment of the activity than SRT participants.
3. MBTS will result in greater pre- to post-intervention increases in positive affect and decreases in anxiety as measured as compared to the SRT participants.
4. MBTS participants will exhibit improved outcomes, as compared to the SRT group, in the 3-month post-intervention period.

ELIGIBILITY:
Inclusion Criteria:

* At least one psychiatric or substance use disorder
* At least one Mental Health Service appointment within the previous 12 months

Exclusion Criteria:

* Active psychosis
* Significant cognitive impairment and/or physical impairment that would preclude participation in the activities
* Previous participation in a therapeutic sailing intervention offered by the VA Salt Lake City Health Care System.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Difference in the change of Acceptance and Action Questionnaire (AAQ2) measure for MBTS and SRT | through study completion, an average of 3 years
  We want to determine if MBTS will result in greater pre- to post-intervention increases in psychological flexibility, as measured by the Acceptance and Action Questionnaire (AAQ2), than a standard recreation therapy activity (SRT). The scale for each question of AAQ2 ranges from 1 to 7. A larger score means a worse outcome-less flexibility.
Difference in the change of Toronto Mindfulness Scale (TMS) measure for MBTS and SRT | through study completion, an average of 3 years
  We want to determine if MBTS will result in greater pre- to post-intervention increases in state mindfulness, as measured by the Toronto Mindfulness Scale (TMS), than a standard recreation therapy activity (SRT). The scale for each question of TMS ranges from 0 to 4. A larger score means a better outcome-greater curiosity or decentering depending on the question.
Difference in the change of Positive and Negative Affect Scale (PANAS)measure for MBTS and SRT | through study completion, an average of 3 years
  We want to determine if MBTS will result in greater pre- to post-intervention increases in positive affect, as measured by the Positive and Negative Affect Scale (PANAS), as compared to the SRT participants. The scale for each question of PANAS ranges from 1 to 5. A larger score indicates a positive or negative effect depending on the question.
Difference in the change of State-Trait Anxiety Inventory (STAI) measure for MBTS and SRT | through study completion, an average of 3 years
  We want to determine if MBTS will result in greater pre- to post-intervention decreases in anxiety, as measured by the Spielberger State-Trait Anxiety Inventory (STAI), as compared to the SRT participants. The scale for each question of STAI ranges from 1 to 4. A larger score may indicate greater or smaller level of anxiety depending on a question.
Difference in the change of psychiatric hospitalizations for MBTS and SRT | through study completion, an average of 3 years
  We want to determine if MBTS participants will exhibit improved outcomes, as compared to the SRT group, in the 3 month post-intervention period as measured by number of psychiatric hospitalizations.
Difference in the change of Emergency Department (ED) visits for MBTS and SRT | through study completion, an average of 3 years
  We want to determine if MBTS participants will exhibit improved outcomes, as compared to the SRT group, in the 3 month post-intervention period as measured by number of ED visits for psychiatric reasons.
Difference in the change of Physical Activity Enjoyment Scale (PACES)measure for MBTS and SRT | through study completion, an average of 3 years
  We want to determine if MBTS participants will experience greater enjoyment of the activity, as measured by the Physical Activity Enjoyment Scale (PACES), than SRT participants. The scale for each question of PACES ranges from 1 to 7. A larger score indicates a positive or negative experience with the activity depending on the question.

CONTACTS AND LOCATIONS:
Overall Officials: William R Marchand, MD, Principal Investigator — Salt Lake City Veterans' Administration Medical Center
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No